

## Statistical Analysis Plan

**Sponsor Protocol Number: ACH-CYT-07** 

A Phase I Open Label, Randomized, Two-Way Crossover Study in Healthy Smokers to Investigate the Effect of Food on the Bioavailability of Cytisine in a New Formulation



Version date: 10 July 2018 



Achieve Life Sciences, Inc.: ACH-CYT-07
Statistical Analysis Plan

## Statistical Analysis Plan

Sponsor Protocol Number: ACH-CYT-07

A Phase I Open Label, Randomized, Two-Way Crossover Study in Healthy Smokers to Investigate the Effect of Food on the Bioavailability of Cytisine in a New Formulation

Simbec Protocol ID: RD 735/33914

Author:

Kerry Williams

Version:

Final 1.0

The undersigned have reviewed and revised this SAP and find it to be consistent with the study requirements:



# **TABLE OF CONTENTS**

| 1 | INTRO | DDUCTION | 7 |
|---|---|---|---|
| | 1.1 | GENERAL | 7 |
| | 1.2 | CHANGES FROM PROTOCOL | 7 |
| | 1.3 | CHANGES FROM PREVIOUS VERSIONS OF THE SAP | 7 |
| 2 | STUD | Y OBJECTIVES | 7 |
| 3 | STUD | Y DESIGN | 8 |
| | 3.1 | OVERVIEW | 8 |
| | 3.2 | INCLUSION AND EXCLUSION CRITERIA | 8 |
| | 3.3 | STUDY TREATMENT | 9 |
| | 3.4 | SCHEDULE OF STUDY PROCEDURES | 9 |
| | 3.5 | SAMPLE SIZE CONSIDERATIONS | 10 |
| | 3.6 | RANDOMISATION | 10 |
| 4 | STUD | Y VARIABLES AND COVARIATES | 11 |
| | <b>4.</b> I | PRIMARY VARIABLES | 11 |
| | 4.2 | SECONDARY VARIABLES | 11 |
| 5 | DEFIN | IITIONS AND DERIVED VARIABLES | 12 |
| 6 ANALYSIS SETS | | YSIS SETS | 12 |
| | 6. l | SAFETY SET | 12 |
| | 6.2 | PK SET | 12 |
| | 6.3 | URINE EXCRETION SET | 13 |
| 7 | SAFE | TY MONITORING | 13 |
| 8 | INTER | RIM ANALYSES | 13 |
| 9 | DATA | | 13 |
| | 9.1 | CRF DATA | 13 |
| | 9.1.1 | Laboratory Data | 13 |
| | 9.1.2 | Pharmacokinetic Data | |
| | 9.2 | RANDOMISATION LIST | |
| | 9.3 | PROGRAMMING AND DATA REVIEW | 14 |
| 10 | STATI | ISTICAL METHODS | |
| | 10.1 | GENERAL PRINCIPLES | |
| | 10.2 | STRATIFICATION AND COVARIATE ADJUSTMENT | |
| | 10.3 | MISSING DATA | |
| | 10.4 | POOLING OF SITES | |
| | 10.5 | MULTIPLE COMPARISONS | 16 |

| | 10.6 | SUBGROUP ANALYSES | 16 |
|----|--------|------------------------------------------|------|
| | 10.7 | STATISTICAL ISSUES | 16 |
| 11 | STATIS | STICAL OUTPUT | .16 |
| | 11.1 | SUBJECT DISPOSITION | . 16 |
| | 11.2 | SUBJECT CHARACTERISTICS AT BASELINE | . 17 |
| | 11.2.1 | Demographic and Baseline Characteristics | . 17 |
| | 11.3 | EFFICACY ANALYSES | . 17 |
| | 11.4 | PK ANALYSES | . 17 |
| | 11.4.1 | Plasma Concentration Data | . 17 |
| | 11.4.2 | Derived Plasma PK Parameters | . 18 |
| | 11.4.3 | Urine Concentration Data | 20 |
| | 11.4.4 | Derived Urine PK Parameters | 20 |
| | 11.5 | PD ANALYSES | 21 |
| | 11.6 | SAFETY ANALYSES | 21 |
| | 11.6.1 | Adverse Events | 21 |
| | 11.6.2 | Laboratory Data | 22 |
| | 11.6.3 | Vital Signs | 23 |
| | 11.6.4 | Electrocardiogram | 23 |
| | 11.7 | OTHER DATA | 23 |
| | 11.7.1 | Prior and Concomitant Medications | 23 |
| | 11.7.2 | All Other Data | 23 |
| 12 | VALID | ATION | 24 |
| 13 | LITERA | ATURE CITATIONS/REFERENCES | 24 |
| 14 | LIST O | F TABLES, FIGURES AND LISTINGS | 25 |
| 15 | SHELL | S FOR TABLES, FIGURES AND LISTINGS | 30 |
| 16 | APPEN | IDICES | 88 |
| | 16.1 | NORMAL RANGES | 88 |



| ADaM | Analysis Data Model |
|---|---|
| AE | Adverse Event |
| Ae | Amount Excreted |
| ANOVA | Analysis of Variance |
| AUC | Area Under the Plasma Concentration Curve |
| AUC <sub>0-∞</sub> | Area Under the Plasma Concentration-time Curve calculated from the time of dosing to infinity |
| $AUC_{0\text{-}t}$ | Area Under the Plasma Concentration-time Curve calculated from the time of dosing to the last measurable concentration |
| BLQ | Below Limit of Quantification |
| BMI | Body Mass Index |
| CI | Confidence Interval |
| $C_{\text{max}}$ | Maximum observed plasma concentration |
| CRF | Case Report Form |
| CS | Clinically Significant |
| CSR | Clinical Study Report |
| CumAe | Cumulative Amount Excreted |
| CV | Coefficient of Variation |
| DBL | Database Lock |
| DMP | Data Management Plan |
| DRM | Data Review Meeting |
| ECG | Electrocardiogram |
| GM | Geometric Mean |
| ICH | International Conference on Harmonisation |
| IMP | Investigational Medicinal Product |
| LLOQ | Lower Limit of Quantification |
| LSMean | Least Squares Mean |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligram |
| mL | Millilitre |


# Achieve Life Sciences, Inc.: ACH-CYT-07 Statistical Analysis Plan

| NCS | Not Clinically Significant |
|-----------|---------------------------------------------------------------|
| PD | Pharmacodynamic |
| PK | Pharmacokinetics |
| PT | Preferred Term |
| QC | Quality Control |
| RBC | Red Blood Cell |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SDTM | Study Data Tabulation Model |
| SOC | System Organ Class |
| TEAE | Treatment Emergent Adverse Event |
| TFL | Table/Figure/Listing |
| $T_{max}$ | Time from dosing to the maximum observed plasma concentration |
| ULOQ | Upper Limit of Quantification |
| WBC | White Blood Cell |




## 1 INTRODUCTION

#### 1.1 GENERAL

This statistical analysis plan (SAP) describes the statistical methods to be used during the reporting and analysis of data collected under the ACH-CYT-07 protocol dated 3<sup>rd</sup> April 2018 and should be read in conjunction with the study protocol and case report form (CRF).

This version of the plan has been developed using the protocol version 2.0 dated 3<sup>rd</sup> April 2018 and the annotated CRF. Any further changes to the protocol or CRF will be reviewed for potential impact on the SAP, which will be amended if it is deemed necessary.

Draft versions of the SAP will undergo review by the Statistical Reviewer, Project Manager, PK Analyst, Medical Writer, Principal Investigator and the Sponsor/Sponsor representative. The analysis plan will be finalised and approved by the Sponsor prior to Database Lock (DBL).

#### 1.2 CHANGES FROM PROTOCOL

- Vital signs summary included.
- The definitions of the PK Set and Urine Excretion Set have been amended to align with the ACH-CYT-01 study. Subjects will be required to receive both doses of cytisine in order to be included in the PK/Urine Excretion Set rather than just one dose,
- The PK parameters, CL/F and Vd/F, will also be presented in line with FDA guidance.

#### 1.3 CHANGES FROM PREVIOUS VERSIONS OF THE SAP

Not applicable.

## 2 STUDY OBJECTIVES

This study will evaluate if there is any food effect for cytisine in a new formulation and further define renal elimination of cytisine over 48 hours.

#### **Primary Objective:**

The primary objectives of this study are:

- 1. To compare the bioavailability ( $C_{max}$  and  $AUC_{0-\infty}$ ) of cytisine in smokers under fed and fasted conditions, following administration of 3 mg cytisine (2 x 1.5 mg cytisine tablets).
- 2. To assess the extent of renal elimination (Ae and Ae%) of cytisine via measurement of urinary concentrations, following administration of 3 mg cytisine (2 x 1.5 mg cytisine tablets).

#### **Secondary Objectives:**

The secondary objectives of this study are:

1. To compare the AUC<sub>0-t</sub>,  $T_{1/2}$ , and  $T_{max}$  of cytisine in subjects under fed and fasted conditions, following administration of 3 mg cytisine (2 x 1.5 mg cytisine tablets).




2. To assess the safety and tolerability of cytisine in a new formulation at the 3 mg dose level under fed and fasted conditions.

## 3 STUDY DESIGN

#### 3.1 OVERVIEW

This is an open-label, randomized, 2-period, single-dose crossover Phase I study conducted in I2 healthy smokers to determine the comparative bioavailability and renal elimination of cytisine following single-dose administration under fed and fasted conditions.

Figure 1: Study Design Overview



The study is comprised of a pre-study screen, followed by 2 treatment periods (I and 2) and a post-study follow-up. Screening assessments will be carried out within 28 days prior to first administration of cytisine. Eligible subjects will receive a single dose of cytisine under fed and fasted conditions during 2 treatment periods. Each treatment period will be of approximately 2 days duration in which blood and urine samples will be collected over 48 h period post-cytisine dosing. Subjects will arrive at the Clinical Unit on Day 0 and will undergo an overnight fast of at least 10 h prior to first dosing on Day I. Randomisation will occur on the morning of Day I, Period I, and cytisine will be administered under fasted (after an overnight fast of at least 10 h) or fed (after a high fat breakfast) conditions. Subjects will complete all 48 h post-dose assessments prior to starting Period 2 and the second dosing day on Day 3. A Post-Study telephone follow-up will be conducted 6 to 8 days after the second dose of cytisine.

#### 3.2 INCLUSION AND EXCLUSION CRITERIA

To be eligible for inclusion into this study, each subject must fulfil all inclusion criteria and not violate any exclusion criteria (for the protocol under which they are entered) during screening prior to randomisation. Details of the inclusion and exclusion criteria are presented within the protocol (sections 6.1, 6.2).




#### 3.3 STUDY TREATMENT

Each subject will receive the following over 2 treatment periods in accordance with the randomisation schedule:

- 3 mg Cytisine (2 x 1.5 mg film coated tablets ( under fasted conditions;
- 3 mg Cytisine  $(2 \times 1.5 \text{ mg film coated tablets } (3 \times 1.5 \text{ mg film coated tablets}))$  under fed conditions.

Cytisine should be administered orally in a single dose application of two 1.5 mg tablets taken with 240 mL water.

#### 3.4 SCHEDULE OF STUDY PROCEDURES

| Days | Screening | Baseline | Study Day (Pe | riod | l and | Period | 1 2) | Post-Study<br>Telephone Call |
|---|---|---|---|---|---|---|---|---|
| Days | -28 to -I | Day 0 | ı | 2 | 3 | 4 | 5 | 6-8 days after last<br>dose |
| Written informed consent | Х | | | | | | | |
| Demographic data/height/weight | Х | | | | | | | |
| Randomization | | | X (Pre-first dose in Period 1) | | | | | |
| Vital signs | Х | Х | XI | | Χ¹ | | Х | |
| Medical history | Х | | | | | | | |
| Medical history update | | X <sup>2</sup> | | | | | | |
| Prior and concomitant medication | Х | Х | Х | Х | Х | Х | Х | |
| Physical examination | Х | | | | | | | |
| 12-lead ECG | Х | | | | | | X <sup>3</sup> | |
| Pregnancy test for all females | X (Serum) | X (Urine) | | | | | | |
| FSH (post-menopausal females only) | Х | | | | | | | |
| Haematology | Х | | | | | | Х | |
| Biochemistry | Х | | | | | | Х | |
| Urinalysis | Х | | | | | | Х | |
| Drugs-of-abuse tests in urine | Х | Х | | | | | | |
| Verification of eligibility criteria | Х | Х | Х | | | | | |
| Cytisine administration | | | Х | | Х | | | |
| Blood collection for PK analysis | | | Х | Х | Х | Х | Х | |
| Urine collection for PK analysis | | | Х | Х | Х | Х | Х | |
| Adverse events monitoring | | X <sup>4</sup> | X <sup>4</sup> | X <sup>4</sup> | X <sup>4</sup> | X <sup>4</sup> | X <sup>4</sup> | X <sup>4</sup> |

Vital signs (supine blood pressure, pulse rate and oral temperature) will be recorded at pre-dose and again approximately 2 hours after administration on Day I of each period.


<sup>&</sup>lt;sup>2</sup> Clinically relevant changes will be reported as adverse events.

Repeat 12-lead ECG and assess prior to discharge on Day 5.

<sup>&</sup>lt;sup>4</sup> Adverse event recording to begin upon admissions on Day 0 of Period 1 to post study.



#### 3.5 SAMPLE SIZE CONSIDERATIONS

A total of 12 subjects will be randomized to the study, with 6 subjects per treatment schedule arm.

Subject numbers are based on the following guidance: In study ACH-CYT-01, geometric mean  $AUC_{0-\infty}$  values in the fed and fasted states were 168 ng.h/mL and 173 ng.h/mL respectively (yielding a geometric mean ratio of 0.97) with an intra subject CV% of approximately 6%. Geometric mean  $C_{max}$  values in the fed and fasted states were 22.3 ng/mL and 29.8 ng/mL respectively (yielding a geometric mean ratio of 0.75) with an intra subject CV% of approximately 23%. Although this study is not a formal comparison of bioequivalence the assumptions used for a typical bioequivalence study have been used in order to estimate an appropriate sample size. Based on the assumption that similar results will be observed for this study, a sample size of 4 subjects would be sufficient to detect a 20% difference in  $AUC_{0-\infty}$  between the treatments with a power of 80%, an alpha of 5% and a fed/fasted ratio of 1. Therefore, 12 subjects, which is the minimum number of subjects recommended for this type of trial, should be sufficient to compare the bioavailability with respect to AUC in the fed and fasted states. Given that the  $C_{max}$  geometric mean ratio observed in the previous study did not fall within the bioequivalence range, likely due to the slower rate of absorption in the fed state, the sample size has been based on  $AUC_{0-\infty}$ .

Subjects who withdraw from the study before receiving any study medication will be replaced. Subjects who are withdrawn from the study due to significant drug-related AEs will not be replaced. Replacement of all other subjects withdrawn from the study after receiving study medication will be decided on a case-by-case basis by the Principle Investigator (or delegate) and Sponsor.

#### 3.6 RANDOMISATION

Subjects will be allocated to a treatment schedule (sequence) in accordance with a randomisation code produced by using the PROC PLAN procedure of SAS® version 9.3. Treatment schedules are as follows:

#### **Schedule A (6 subjects):**

- Period I: Cytisine (2 x 1.5 mg tablets) will be administered 30 minutes after the start of a high fat breakfast (fed state) with 240 mL water.
- Period 2: Cytisine (2 x 1.5 mg tablets) will be administered after the overnight fast of at least 10 hours (fasting state with 240 mL water.

### Schedule B (6 subjects):

- Period I: Cytisine (2 x 1.5 mg tablets) will be administered after the overnight fast of at least 10 hours (fasting state with 240 mL water.
- Period 2: Cytisine (2 x 1.5 mg tablets) will be administered 30 minutes after the start of a high fat breakfast (fed state) with 240 mL water.

Subjects will be numbered sequentially from 001 (i.e. 001, 002 etc.). Any replacement subjects will be assigned the same randomisation as the subjects they are replacing with 100 added to the subject number (i.e. 101 would replace 001 etc.).




## 4 STUDY VARIABLES AND COVARIATES

### 4.1 PRIMARY VARIABLES

The primary plasma cytisine pharmacokinetic endpoints for this study are as follows:

• C<sub>max</sub> Maximum observed plasma concentration post dose, obtained from the

observed concentration versus time profile.

•  $AUC_{0-\infty}$  Total area under the plasma concentration-time curve (AUC) from zero

to infinity, calculated as  $AUC_{0-\infty} = AUC_{0-t} + (C_{last}/\lambda_z)$ , where  $C_{last}$  is the last measurable plasma concentration and  $\lambda_z$  the apparent terminal

elimination rate constant.

The primary urine cytisine pharmacokinetic endpoints for this study are as follows:

Ae Amount excreted in urine over time.

Ae% Percentage of drug excreted in urine.

## 4.2 SECONDARY VARIABLES

The secondary plasma cytisine pharmacokinetic endpoints for this study are as follows:

• T<sub>max</sub> Time of occurrence of maximum observed plasma concentration.

 $\bullet$  AUC<sub>0-t</sub> AUC from the time of zero to the last sampling time at which

concentrations were at or above the lower limit of quantification (LLOQ),

calculated by the linear-up/log-down trapezoidal rule.

• %AUC Residual area or percentage of extrapolated part for the calculation of

 $AUC_{0-\infty}$ , calculated as  $100*[1-(AUC_{0-t}/AUC_{0-\infty})]$ .

•  $\lambda_z$  Apparent terminal elimination rate constant.

•  $t_{1/2}$  Apparent terminal elimination half-life, calculated from  $\ln 2/\lambda_z$ .

CL/F Apparent total body clearance.

Vd/F
 Apparent volume of distribution.

The safety endpoints for this study are as follows:

- Adverse events (AEs).
- Laboratory safety data (biochemistry, haematology, urinalysis and microscopy).
- Vital signs (supine systolic/diastolic blood pressure, pulse rate and oral temperature).
- 12-lead ECG (heart rate, PR interval, QRS width, QT interval and QT interval corrected using Fridericia's formula (QTcF interval)).




## 5 DEFINITIONS AND DERIVED VARIABLES

**Study drug/IMP:** Study drug/IMP means 3 mg cytisine (2 x 1.5 mg cytisine tablets).

**Treatment:** Treatment means 3 mg cytisine in the fed or fasted state.

**Baseline:** In general, baseline is defined by subject and by variable as the last non-missing value (including repeats) before the first dose of study drug. This is normally the pre-dose assessment on Day I but if this assessment is missing (or not planned) then the assessment at the Screening/Day 0 visit will be used instead if available.

**Study Day**: Study day is the number of days since start of treatment where the date of first dose is counted as Day I.

**Bleed Time Deviation:** Actual time of blood sample – theoretical time of blood sample.

**Protocol Deviation:** a deviation related to study inclusion or exclusion criteria, conduct of the trial, subject management or subject assessment. This refers to any change, divergence, or departure from the study design or procedures defined in the protocol. Deviations recorded by the Project Manager or detected by Data Management or by statistical programming checks will be identified and discussed at the Data Review Meeting (DRM) before Database Lock (DBL). All protocol deviations within the study database will be classified as either 'Major' or 'Minor' prior to DBL, details of which will be included within the Protocol Deviations listing.

## **6 ANALYSIS SETS**

Membership of the analysis sets will be reviewed and agreed prior to DBL. These will be reviewed by the Sponsor, Study Statistician, PK analyst and Project Manager and signed off. If PK data is not available at the time of DBL, then subjects will be assumed to be included in the analysis set unless the PK data provide reason to exclude a subject, in which case this will be discussed with the Sponsor and documented within the Analysis Sets listing (Listing 16.2.3.1).

#### **6.1 SAFETY SET**

All randomised subjects who receive at least one dose of cytisine will constitute the Safety Set.

This analysis set will be used for baseline and safety summaries as well as for all study listings.

#### 6.2 PK SET

The PK Set will include all subjects who receive both doses of cytisine and have sufficient plasma concentration-time profiles complying with the following criteria:

- Do not have an occurrence of vomiting or diarrhoea which renders the concentration profile unreliable (e.g. if vomiting occurs at or before 2 times median  $T_{max}$ );
- Do not use a concomitant medication which renders the concentration profile unreliable;
- Do not have a pre-dose concentration that is greater than 5% of the corresponding C<sub>max</sub>;


- Have at least one evaluable concentration that is preceded by a lower evaluable concentration and followed by a lower evaluable concentration for the calculation of C<sub>max</sub>, T<sub>max</sub> and AUCs (i.e. at least 3 evaluable concentrations in total);
- Do not violate the protocol (major protocol deviation) in a way that may invalidate or bias the results.

#### 6.3 URINE EXCRETION SET

The Urine Excretion Set will include all subjects who receive both doses of cytisine and have sufficient urine excretion profiles complying with the following criteria:

- Do not have any missing urine excretion collections (i.e. missing urine in a collection period specified in section 1.4.3) which renders analysis of overall excretion unreliable;
- Do not have an occurrence of vomiting or diarrhoea which renders the urine excretion profile unreliable (e.g. if vomiting occurs at or before 2 times median T<sub>max</sub> derived from plasma data);
- Do not use a concomitant medication which renders the concentration profile unreliable;
- Do not violate the protocol (major protocol deviation) in a way that may invalidate or bias the results.

## 7 SAFETY MONITORING

No interim safety analyses are planned for this study.

## 8 INTERIM ANALYSES

No interim efficacy/PK analyses are planned for this study.

#### 9 DATA

#### 9.1 CRF DATA

| CRF data will be provided by | Data Management to the Statistics department as SAS datasets in |
|---|---|
| standard format. SDTM datas | ets will be derived from the raw database and ADaM from SDTM. |
| Both SDTM and ADaM domains will be | be used for programming the outputs to be included in the Clinical |
| Study Report (CSR). SDTM/ADaM | programming will begin when populated standard SAS |
| datasets are available. | |

#### 9.1.1 Laboratory Data

Transfers of safety laboratory data will be available from the Pathology laboratory and delivered to Data Management via electronic transfer and stored within the study database. Details of laboratory data are documented in the Data Management Plan (DMP). Populated test transfers will be received before programming can start. The following results will be included:


- Haematology: Haemoglobin, haematocrit, r
  - **Haematology**: Haemoglobin, haematocrit, mean cell volume, mean cell haemoglobin, mean cell haemoglobin concentration, red blood cells, white blood cells, neutrophils, lymphocytes, monocytes, eosinophils, basophils and platelets.
  - **Biochemistry**: Total protein, albumin, total bilirubin, alanine transaminase, aspartate transaminase, gamma glutamyl transferase, alkaline phosphatase, glucose, sodium, potassium, calcium, bicarbonate, creatinine and urea.
  - **Urinalysis:** Glucose, specific gravity, protein, leucocytes, ketones, urobilinogen, bilirubin, nitrites, pH and blood.
  - **Microscopy:** In the event that the 'dipstick' is positive, RBCs, WBCs, epithelial cells, crystals, bacteria and casts will be examined microscopically.
  - Virology: Hep B, Hep C and HIV.
  - **Drugs of Abuse and Alcohol:** Urine alcohol and drugs of abuse screen: cannabinoids, amphetamines, cocaine, benzodiazepines, opiates and cotinine.
  - **Pregnancy/post-menopausal assessment:** serum/urine pregnancy test and follicle stimulating hormone.
  - Other parameters: Any further parameters that are taken that are not included as part of the above categories will be included in an 'Other Laboratory Data' listing.

#### 9.1.2 Pharmacokinetic Data

Plasma and urine concentration data will be received as an Excel file from the Bioanalytical department via an electronic transfer and stored as a SAS dataset. This data will then be stored in the appropriate SDTM domain and subsequent ADaM domain which will be used to produce the file provided to the pharmacokinetic team in order to derive the PK parameters using Phoenix WinNonlin 6.4. Derived PK parameters will be received by the Statistics department from the Project Manager/PK analyst in a SAS.xpt file in an agreed format and then stored as a SAS dataset and subsequently within SDTM/ADaM domains.

#### 9.2 RANDOMISATION LIST

The randomisation list will be uploaded to a SAS dataset and incorporated into the relevant SDTM/ADaM domains.

#### 9.3 PROGRAMMING AND DATA REVIEW

Programming of datasets, tables, figures and listings may be ongoing while study data management activities are in progress.

Prior to DBL, a review of the clinical database (i.e. CRF data, laboratory data) in the form of Excel data listings will be conducted. A Data Review Meeting (DRM) will be held to discuss the outcome of this review, any potential impact on the analyses, analysis sets and protocol deviations. Once all data issues have been resolved and the analysis sets approved, the database will be locked. The SDTM/ADaM datasets will be finalised and the final run of outputs and quality control (QC) will take place.




## 10 STATISTICAL METHODS

#### 10.1 GENERAL PRINCIPLES

- All statistical methods will be based on the International Conference on Harmonisation (ICH)
   E9 document "Statistical Principles for Clinical Trials".
- All data collected will be presented within data listings and any unscheduled visits will be listed.
- Data will be summarised by treatment and overall (data from both treatments pooled) where appropriate. The format of the summaries is defined in the shells at the end of this document.
- In summary and analysis tables of continuous variables, standard descriptive statistics (N [number within population], n [number of observations included in analysis], mean, standard deviation [SD], median, minimum and maximum) will be presented. Least squares mean (LS mean) and 90/95% confidence interval (CI) will be presented in the statistical analysis outputs as appropriate. For PK summaries, geometric mean, and coefficient of variation (%CV) will also be used to summarise the data.
- Unless otherwise specified, the minimum and maximum statistics will be presented in summary tables to the same number of decimal places as the original data. The mean, median, LS mean, geometric mean and CI will be presented to one more decimal place than the original data. SD will be presented to two more decimal places than the original data. %CV will be presented to one decimal place.
- In summary tables of categorical variables, the number of non-missing observations by category
  will be presented along with percentages. Unless otherwise specified, the denominator for each
  percentage will be the number of non-missing observations. All percentages will be presented
  to one decimal place.
- All plots will use a linear time scale for the nominal times of the visits and will be labelled by time point.
- Original values will be used in summary tables, unscheduled measurements will be listed only.
  However, where repeats of baseline values occur, the last assessment will be used within any
  summary tables and used to calculate change from baseline. In case an unscheduled measurement
  is performed immediately after the scheduled measurement due to an error in the original
  measurement, the unscheduled measurement will be included in the analysis and the original
  erroneous measurement will be excluded.
- The date format for all output presentations will be as captured in the database.
- All statistical analysis will be performed using SAS 9.3 or higher.
- All hypothesis testing will be carried out at the 5% (2-sided) significance level unless stated otherwise.
- P-values will be rounded to four decimal places. P-values less than 0.0001 will be reported as
   <0.0001 in tables.</li>
- Generally, character values will be left aligned and numeric values will be decimally aligned.
- If any of the assumptions underlying the formal statistical methods proposed are violated during
  the analysis of the final data, alternative statistical methods will be used and any changes
  documented in the statistical methods section of the clinical study report (CSR), including the
  rationale for use.


Statistical Analysis Plan

- For numeric data which includes non-numeric values (e.g. PK data reported as BLQ or laboratory results reported as < 10 or >100) the following principles will be applied when summarising the data:
  - > BLQ will be replaced with a zero.
  - Results reported as <x or >x will be treated as x.

#### 10.2 STRATIFICATION AND COVARIATE ADJUSTMENT

Not applicable.

#### 10.3 MISSING DATA

Generally, no methods to impute missing data will be used. However, for the purpose of calculating change from baseline, in the instance of a missing baseline result for Period I (generally the assessment at Day I, Pre-Dose) the results obtained at the Screening/Day 0 visit will be used instead, if available. Missing Period 2 baseline results will not be replaced.

In the instance of missing pharmacokinetic blood samples, the linear trapezoidal rule will be employed between the samples immediately before and after the missing sample for the AUC calculations.

#### 10.4 POOLING OF SITES

Not applicable.

#### 10.5 MULTIPLE COMPARISONS

Not applicable.

### 10.6 SUBGROUP ANALYSES

Not applicable.

#### 10.7 STATISTICAL ISSUES

None.

## 11 STATISTICAL OUTPUT

General principles for layout of the statistical output are described in Section 10.1. Layout and specifications are illustrated for each unique table and listing within the shells presented in Section 14.

#### 11.1 SUBJECT DISPOSITION

The subject disposition table will summarise the following data for all randomised subjects:


Statistical Analysis Plan

- The number (%) of subjects within each analysis set;
- The number (%) of subjects receiving each treatment;
- The number (%) of subjects within each treatment schedule (sequence);
- The number (%) of subjects who completed each study period, where completion is defined as having the 48 h sample collections on Day 3 (Period I) or Day 5 (Period 2).
- The number (%) of subjects who completed the study/withdrew from the study and the associated reasons for early study termination. A subject is deemed to have completed the study if they complete the Post-Study follow-up telephone contact.

Screening and study completion/termination data will also be listed. A listing of all subjects with protocol deviations will be presented including major/minor classification. A data listing presenting subject eligibility for each analysis set and the reason for exclusion from an analysis set will also be presented.

#### 11.2 SUBJECT CHARACTERISTICS AT BASELINE

#### 11.2.1 Demographic and Baseline Characteristics

Demographic data will be listed (including informed consent information) and descriptive statistics for the continuous variables age, height, weight and BMI and frequencies for the categorical variable race will be tabulated by gender and overall.

Demographic and baseline data will be listed and summarised using the Safety Set. Demographic data may also be summarised using the PK Set/Urine Excretion Set, if appropriate.

### 11.3 EFFICACY ANALYSES

Not applicable.

### 11.4 PK ANALYSES

The primary analysis sets for summaries of plasma and urine PK data will be the PK Set and Urine Excretion Set respectively. If the PK Set/Urine Excretion Set and the Safety Set are not equivalent, then all PK summaries described below will also be produced for the Safety Set.

#### 11.4.1 Plasma Concentration Data

Plasma PK samples will be collected for measurement of cytisine at the following time points during each period: Pre-dose, 15 min, 20 min, 30 min, 45 min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h, 14h, 16h, 24h and 48h post-dose.

Cytisine concentrations in plasma will be listed and summarised for each treatment using the descriptive statistics N, n, arithmetic mean, arithmetic standard deviation (SD), coefficient of variation (CV%), minimum, median and maximum.

The individual subject plasma cytisine concentration profiles over time will be presented graphically using actual blood sampling times on a linear and semi-logarithmic scale for each subject with both treatments


presented on the same plot. Arithmetic mean plasma cytisine concentration profiles over time will be presented on linear and semi-logarithmic scales.

For inclusion within the summary tables and linear scale plots, concentrations below the limit of quantification (BLQ) will be assigned a value of zero. Concentrations above the upper limit of quantification (ULOQ) will be obtained via dilution into the calibration range and are valid results. For inclusion within the semi-logarithmic scale plots, concentrations below the limit of quantification will be set to missing.

Plasma concentration data listings and individual plots will be presented using the Safety Set. Plasma concentration data summaries and mean plots will be presented using the PK Set and also the Safety Set if it differs from the PK Set. All plasma concentration data included in listings and summaries will be presented to three significant figures.

#### 11.4.2 Derived Plasma PK Parameters

The following derived pharmacokinetic parameters of cytisine in plasma will be determined using WinNonlin Phoenix 6.4 from the individual concentration versus time profiles using standard non-compartmental methods:

| Pharmacokinetic<br>Parameter | Definition | WinNonlin computation | WinNonlin<br>Parameter<br>Name |
|---|---|---|---|
| C <sub>max</sub> (ng/mL) | Maximum observed plasma concentration post dose | Maximum observed concentration, occurring at Tmax. If not unique, then the first maximum is used. | Cmax |
| T <sub>max</sub> (h) | Time of occurrence of maximum observed plasma concentration | Time of maximum observed concentration. If the maximum observed concentration is not unique, then the first maximum is used. | Tmax |
| AUC <sub>0-t</sub> (h*ng/mL) | The area under the plasma concentration-time curve (AUC) from 0 h to the last sampling time at which concentrations were at or above the LLOQ | AUC measured from the concentration at time of dosing to the last measurable positive concentration. The AUC is computed using the linear-up/log-down trapezoidal method. | AUClast |
| AUC <sub>(0-inf)</sub> (h*ng/mL) | The AUC from 0 h extrapolated to infinity | AUC measured from the concentration at time of dosing extrapolated to infinity based on the last observed concentration. $= AUC_{0-t} + \frac{C_{lastobs}}{\lambda_z}$ | AUCINF_obs |
| AUC <sub>% extrapolated</sub> (%) | Residual area. | Percentage of AUC <sub>0-inf</sub> due to extrapolation from time of last measurable positive concentration to infinity. $= \frac{AUC_{0-inf} - AUC_{0-t}}{AUC_{0-inf}} \cdot 100$ | AUC_%Extrap_<br>obs |
| λ <sub>z</sub> (1/h) | Apparent terminal elimination rate constant. | First order rate constant associated with the terminal (log-linear) | Lambda_z |


| | | portion of the curve. Estimated by linear regression of time vs. log concentration; the regression analysis should contain data from at least 3 different time points in the terminal phase. | |
|---|---|---|---|
| t <sub>1/2</sub> (h) | Apparent terminal elimination half-life. | $=\ln(2)/\lambda_z$ | HL_Lambda_z |
| CL/F | Apparent total body clearance. | $= Dose/AUC_{0-inf}$ | Cl_F_obs |
| Vd/F | Apparent volume of distribution based on the terminal phase. | $= \frac{Dose}{K_{el}.AUC_{0-inf}}$ | Vz_F_obs |

The terminal elimination rate constant  $(\lambda_z)$  will be determined by plotting the concentration data versus time on a semi-logarithmic scale. The parameter will be estimated by linear least square regression analysis, using the last three (or more) non-zero concentrations. The upper and the lower time points, as well as the number of time points, used for  $\lambda_z$  estimation will be reported. Values of  $\lambda_z$ , AUC<sub>0...</sub>, %AUC and  $t_{1/2}$  will not be reported for cases where  $\lambda_z$  cannot be reliably determined.

AUC<sub>0-t</sub> will be calculated using the linear-up/log-down trapezoidal method.

For the calculation of derived pharmacokinetic parameters, concentrations below the limit of quantification (BLQ) will be assigned a value of zero. In case of a deviation from the theoretical time, the actual time of blood sample will be used in the calculation of the derived pharmacokinetic parameters. Should the actual time be unavailable but a blood sample was taken, the nominal time point will be assigned.

Derived pharmacokinetic parameters will be listed and summarised for each treatment. The descriptive statistics presented will be N, n, arithmetic mean, arithmetic standard deviation (SD), coefficient of variation (CV%), minimum, median, maximum and geometric mean (with the exception of  $T_{max}$ ).

If no reliable PK parameter can be determined for more than a third of the subjects, only n, minimum and maximum values will be presented for that parameter and all other descriptive statistics will be omitted.

Plasma PK parameter data listings will be presented using the Safety Set. Plasma PK data summaries will be presented using the PK Set and also the Safety Set if they differ. All PK parameter data included in listings and summaries will be presented to three significant figures with the exception of the CV% which will be presented to one decimal place.

#### 11.4.2.1 Statistical Analysis of Plasma PK Parameters

Following logarithmic transformation,  $C_{max}$ ,  $AUC_{0-t}$ , and  $AUC_{0-w}$  values will be subjected to an analysis of variance (ANOVA) including fixed effects for sequence (treatment schedule), period, treatment and subject nested within sequence. Point estimates and 90% confidence intervals (CI) will be constructed for the contrasts between fed and fasted states using the residual mean square error obtained from the ANOVA. The point and interval estimates will be back-transformed to give estimates of the ratios of the geometric least squares means (LSmean) and corresponding 90% CI. In addition, estimated geometric means will be presented.




A comparison of  $T_{\text{max}}$  will be performed using the Wilcoxon Signed-Rank test. In addition, the Hodges-Lehmann estimate of the median difference in  $T_{\text{max}}$  and 95% CI will be presented.

The statistical analysis of the plasma PK parameters will be performed using the PK Set and also the Safety Set if they differ. Geometric LSmeans will be presented to three significant figures and the ratios and 90% Cls will be presented to 2 decimal places.

#### 11.4.3 Urine Concentration Data

Urine PK samples will be collected for measurement of cytisine at the following time intervals during each study period: Pre-dose, 0-2h, 2-4h, 4-8h, 8-12h, 12-24h, 24-26h, 26-28h, 28-32h, 32-36h, 36-48h post-dose.

Cytisine concentrations in urine will be listed and summarised for each using the descriptive statistics N, n, arithmetic mean, arithmetic standard deviation (SD), coefficient of variation (CV%), minimum, median and maximum.

Urine concentrations will be listed using the Safety Set and summarised using the Urine Excretion Set. The summary may also be presented using the Safety Set if it differs from the Urine Excretion Set. All urine concentration data included in listings and summaries will be presented to three significant figures.

#### 11.4.4 Derived Urine PK Parameters

The derived urine pharmacokinetic parameters, Ae and Ae% (individual and cumulative), will be determined from the individual concentration versus time data using SAS version 9.3.

The derived urine PK parameter Ae will be calculated as: urine volume \* urine cytisine concentration. Ae% will be derived as: 100\*Ae/Dose (where dose is expressed in ng). The cumulative parameters (CumAe, CumAe%) are the sum of the individual values calculated for each time interval from 0h to 48h. Total  $Ae_{0.48h}$  is defined as the total amount excreted from 0 h to 48 h.

For the calculation of derived urine pharmacokinetic parameters, concentrations below the limit of quantification will be assigned a value of zero.

The derived urine parameters Ae, Ae%, CumAe and CumAe% for each time interval will be listed and summarised with the urine cytsisine concentration data,

The derived urine pharmacokinetic parameters Total Ae<sub>0-48h</sub> and Total Ae<sub>0-48h</sub>% will be listed and summarised separately using the descriptive statistics N, n, arithmetic mean, arithmetic standard deviation (SD), coefficient of variation (CV%), minimum, median, maximum and geometric mean.

Urine PK parameter data listings will be presented using the Safety Set. Urine PK data summaries will be presented using the Urine Excretion Set and also the Safety Set should they differ. Urine PK parameter data included in listings and summaries will be presented to three significant figures with the exception of Ae% and CumAe% which will be presented to one decimal place.




### 11.4.4.1 Statistical Analysis of Urine PK Parameters

Following logarithmic transformation, Total  $Ae_{0-48h}$  values will be subjected to an analysis of variance (ANOVA) including fixed effects for sequence (treatment schedule), period, treatment and subject nested within sequence. Point estimates and 90% confidence intervals (CI) will be constructed for the contrasts between fed and fasted states using the residual mean square error obtained from the ANOVA. The point and interval estimates will be back-transformed to give estimates of the ratios of the geometric least squares means (LSmean) and corresponding 90% CI. In addition, estimated geometric means will be presented.

The statistical analysis of the urine PK parameter will be performed using the Urine Excretion Set and also the Safety Set should they differ. Geometric LSmeans will be presented to three significant figures and the ratios and 90% Cls will be presented to 2 decimal places.

#### 11.5 PDANALYSES

Not applicable.

#### 11.6 SAFETY ANALYSES

#### 11.6.1 Adverse Events

All AEs will be coded using the MedDRA dictionary using the version specified in the Data Management Plan (DMP).

All AEs, including those which occurred prior to the first dose of study drug, will be listed. Only treatment emergent adverse events (TEAEs), i.e., existing conditions that worsen or events that occur during the course of the study after administration of IMP, will be included within the summary tables. AEs occurring post-dose on Period I up to immediately prior to dosing on Period 2 will be assigned to the corresponding Period I treatment. Similarly, any AEs occurring post-dose on Period 2 up to Post-Study will be assigned to the corresponding Period 2 treatment. TEAEs will be summarised by treatment and overall.

An overall summary of AEs will be produced including the number of TEAEs; the number and % of subjects reporting at least I TEAE, serious TEAE (where SAE is reported as 'Yes'), TEAE leading to withdrawal from study drug (Action recorded as 'Study Drug Discontinued'); the number and % of subjects reporting TEAEs by severity and relationship to study drug. A subject with multiple occurrences of any AE is counted only once at the maximum level of severity or the highest association to study drug.

The number of TEAEs and the number and % of subjects reporting at least one TEAE will be tabulated by system organ class (SOC) and preferred term (PT). A subject reporting multiple episodes of a particular AE within a treatment period will only contribute one count towards the corresponding SOC and preferred term. The number of TEAEs and the number and % of subjects reporting at least one TEAE will also be tabulated by preferred term (PT), with the PTs sorted in descending order of frequency. A subject reporting multiple episodes of a particular AE within a treatment period will only contribute one count towards the corresponding PT.


In addition, the number and % of subjects reporting TEAEs will be tabulated by maximum severity and strongest relationship to study drug. For the summary of TEAEs by severity, if a subject has multiple events occurring within the same SOC or preferred term the event with the highest severity will be counted. Similarly, for TEAEs by relationship to study drug, if a subject has multiple events occurring within the same SOC or PT, the event with the highest association to study drug will be counted.

Data will be listed by treatment. For any adverse event taken prior to first administration of study drug, treatment will be described as 'Prior to Treatment'.

Where there are only partial dates/times recorded for adverse events, adverse events will be assigned to treatment unless it can be ruled out based on the partial information.

The derived variables, 'Time from Dose' and 'Duration' will be presented where full date and time are present. If partial dates are present for any parameter required in the calculation, then the variable will not be populated. The following will be used to calculate the variables:

**Duration**: (Date/Time of Resolution-Date/Time of Onset) + 1 minute;

**Time from Dose**: (Date/Time of Onset-Date/Time of Start of Dose).

The following will be presented in listing format within the data summaries:

Serious Adverse Events – If there are none present, the listing will be produced stating: 'No subjects experienced any serious adverse events'.

Adverse Events which Led to Withdrawal of Study Drug – If there are none present, the listing will be produced stating: 'No subjects experienced any adverse events that led to withdrawal of study drug'.

Adverse event data will be summarised and listed using the Safety Set.

#### 11.6.2 Laboratory Data

Routine safety laboratory tests will be carried out at Screening and Day 5.

The safety laboratory parameters required for this study are listed in section 9.1.1.

Safety laboratory data listings will be presented in two ways:

- Out of range values any values that fall outside of the normal/alert ranges (presented in listing format within the data summaries)
- All safety laboratory data (including physician's review (Normal, Abnormal-NCS, Abnormal-CS))
   with any out of range values flagged (presented within the data listings).

Microscopy, virology, urine drugs of abuse and alcohol screen, pregnancy tests and other parameters will also be listed.

If there are no further parameters databased other than those specified in section 9.1.1 then the 'Other Laboratory Data' listings should display, 'No other laboratory parameters to report'.

Laboratory data will be listed using the Safety Set.




#### 11.6.3 Vital Signs

Vital signs will be taken at Screening; Day 0; Day 1 at pre-dose and 2h post-dose (Period 1); Day 3 at pre-dose and 2h post-dose (Period 2); Day 5.

Vital signs parameters (supine systolic and diastolic blood pressure and pulse rate and oral temperature) will be listed with any out of normal range values (see Appendix 16.1) flagged (flag 'H' or 'L' appended to relevant result). Descriptive statistics (N, n, mean, SD, minimum, median and maximum) of absolute and change from pre-dose to 2 h post-dose will be tabulated by treatment.

Vital signs data will be listed and summarised using the Safety Set.

## 11.6.4 Electrocardiogram

#### 11.6.4.1 12-Lead ECG

12-lead ECGs will be performed in triplicate at Screening and prior to discharge on Day 5.

12-lead ECG parameters (heart rate, PR interval, QRS width, QT interval and QTcF interval) will be listed with any out of normal range values (see Appendix 16.1) flagged (flag 'H' or 'L' appended to relevant result). The ECG results will also be assessed as either 'normal' or abnormal' with comments on abnormal results also presented.

12-lead ECG data will be listed using the Safety Set.

### 11.7 OTHER DATA

#### 11.7.1 Prior and Concomitant Medications

All medications will be coded using the WHO Drug Dictionary (version as specified in the DMP) and listed using the ATC Level 4 class, Preferred Term and verbatim text. A medication will be regarded as prior if it stops prior to administration of first treatment and will be assigned a treatment phase of 'Prior to treatment'. A medication which starts prior to first treatment and continues after dosing and will be assigned a treatment phase of 'Prior and ongoing'. Otherwise, treatment phase will be described as the treatment the medication started on. Where there are only partial dates/times recorded for medications, medications will be assigned to all treatments that cannot be ruled out based on the partial information.

Prior and concomitant medications will be listed using the Safety Set.

#### 11.7.2 All Other Data

All data will be listed using the Safety Set, including the following: Tobacco and Alcohol Use, Visit Dates, Medical History, Menstrual and Obstetric History, Physical Examination, Inclusion/Exclusion Criteria Failures, Bag Search and Cigarette Collection, Eligibility Check, Dose Administration and Additional Notes.




### **Derivations within listings:**

<u>PK Blood Sampling Time Deviations</u>: Calculate sample time deviation as: actual time – theoretical time, display in minutes.

<u>Analysis Sets</u>: Detail whether subject should be included in each of the analysis sets along with corresponding comments if not included.

<u>Inclusion/Exclusion Criteria</u>: Only failures to be recorded. If no failures display 'All subjects passed inclusion/exclusion criteria'.

<u>Protocol Deviations</u>: Major/minor classification to be assigned and confirmed by Sponsor.

## 12 VALIDATION

All tables, figures and listings will be subject to independent quality control and visual review. Unique tables will be independently programmed. Findings will be documented in an Output Summary file quality control form and actions taken will also be documented.

## 13 LITERATURE CITATIONS/REFERENCES

None.


# 14 LIST OF TABLES, FIGURES AND LISTINGS

## List of Tables and Figures Contained in Report Section 14

## 14.1 Disposition and Demographic Data

## 14.1.1 Disposition Data

| Table 14.1.1.1 | Summary of Study Disposition | Safety Set |
|----------------|------------------------------|------------|
|----------------|------------------------------|------------|

## 14.1.2 Demographic Data

| Table 14.1.2.1 | Summary of Demographic Data | Safety Set |
|---|---|---|
| Table 14.1.2.2 | Summary of Demographic Data - (if required) | PK Set |
| Table 14.1.2.3 | Summary of Demographic Data - (if required) | Urine Excretion Set |

## 14.2 Efficacy Data

Not Applicable.

## 14.3 Safety Data

## 14.3.1 Adverse Events

| Table 14.3.1.1 | Summary of Treatment Emergent Adverse Events | Safety Set |
|---|---|---|
| Table 14.3.1.2 | Summary of Treatment Emergent Adverse Events by System<br>Organ Class and Preferred Term | Safety Set |
| Table 14.3.1.3 | Summary of Treatment Emergent Adverse Events by Preferred Term | Safety Set |
| Table 14.3.1.4 | Summary of Treatment Emergent Adverse Events by System Organ Class, Preferred Term and Severity | Safety Set |
| Table 14.3.1.5 | Summary of Treatment Emergent Adverse Events by System Organ Class, Preferred Term and Relationship | Safety Set |
| Table 14.3.1.6 | Serious Adverse Events | Safety Set |
| Table 14.3.1.7 | Adverse Events Leading to Withdrawal of Study Drug | Safety Set |

## 14.3.2 Laboratory Safety

| Table 14.3.2.1 | Biochemistry Out of Range Data | Safety Set |
|----------------|--------------------------------|------------|
| Table 14.3.2.2 | Haematology Out of Range Data | Safety Set |
| Table 14.3.2.3 | Urinalysis Out of Range Data | Safety Set |




| Table 14.3.3.1 Post-Dose Vital Signs Data Safety S | Table 14.3.3.1 | Summary of Absolute and Change from Pre-Dose to Post-Dose Vital Signs Data | Safety Set |
|---|---|---|---|
|---|---|---|---|

## **14.4** Pharmacokinetics

## 14.4.1 Concentration-Time Data

| Table 14.4.1.1 | Summary of Plasma Cytisine Concentration Data | PK Set |
|---|---|---|
| Table 14.4.1.2 | Summary of Urine Cytisine Concentration Data | Urine Excretion Set |
| Table 14.4.1.3 | Summary of Plasma Cytisine Concentration Data — (if required) | Safety Set |
| Table 14.4.1.4 | Summary of Urine Cytisine Concentration Data — (if required) | Safety Set |
| Figure 14.4.1.1 | Mean Plasma Cytisine Concentration-Time Curves on a Linear Scale | PK Set |
| Figure 14.4.1.2 | Mean Plasma Cytisine Concentration-Time Curves on a Semi-Logarithmic Scale | PK Set |
| Figure 14.4.1.3 | Mean Plasma Cytisine Concentration-Time Curves on a Linear Scale — (if required) | Safety Set |
| Figure 14.4.1.4 | Mean Plasma Cytisine Concentration-Time Curves on a Semi-<br>Logarithmic Scale — (if required) | Safety Set |

## 14.4.2 Derived Pharmacokinetic Data

| Table 14.4.2.1 | Summary of Derived Plasma Cytisine Pharmacokinetic Parameters | PK Set |
|---|---|---|
| Table 14.4.2.2 | Summary of Derived Urine Cytisine Pharmacokinetic Parameters | Urine Excretion Set |
| Table 14.4.2.3 | Summary of Statistical Analysis of Cytisine $C_{\text{\scriptsize max}}$ and AUC | PK Set |
| Table 14.4.2.4 | Summary of Statistical Analysis of Cytisine $T_{\text{\scriptsize max}}$ | PK Set |
| Table 14.4.2.5 | Summary of Statistical Analysis of Cytisine Total Amount Excreted in Urine | Urine Excretion Set |
| Table 14.4.2.6 | Summary of Derived Plasma Cytisine Pharmacokinetic<br>Parameters — (if required) | Safety Set |
| Table 14.4.2.7 | Summary of Derived Urine Cytisine Pharmacokinetic Parameters – (if required) | Safety Set |
| Table 14.4.2.8 | Summary of Statistical Analysis of Cytisine $C_{\text{max}}$ and AUC – (if required) | Safety Set |
| Table 14.4.2.9 | Summary of Statistical Analysis of Cytisine $T_{max}$ – (if required) | Safety Set |


Table 14.4.2.10 Summary of Statistical Analysis of Cytisine Total Amount Excreted in Urine – (if required)

## 14.5 Pharmacodynamics

Not applicable.

#### 14.6 Other

Not applicable.

## **Subject Data: Listings Contained in Report Appendix 16.2**

## 16.2.1 Visit Dates, Dosing Information and Disposition

| Listing 16.2.1.1 | Visit Dates | Safety Set |
|------------------|---------------------|------------|
| Listing 16.2.1.2 | Dose Administration | Safety Set |
| Listing 16.2.1.3 | Subject Disposition | Safety Set |
| Listing 16.2.1.4 | Additional Notes | Safety Set |

#### 16.2.2 Protocol Deviations

| Listing 16.2.2.1 | Protocol Deviations | Safety Set |
|------------------|---------------------|------------|

## 16.2.3 Analysis Sets

| Listing 16.2.3.1 | Analysis Sets | Safety Set |
|------------------|---------------|------------|

## 16.2.4 Demographic Data and Other Baseline Characteristics

| Listing 16.2.4.1 | Demographic Data | Safety Set |
|-------------------|-------------------------------------------|------------|
| Listing 16.2.4.2 | Medical History and Concurrent Conditions | Safety Set |
| Listing 16.2.4.3 | Virology Results | Safety Set |
| Listing 16.2.4.4 | Tobacco and Alcohol Use | Safety Set |
| Listing 16.2.4.5 | Drugs of Abuse Results | Safety Set |
| Listing 16.2.4.6 | Menstrual and Obstetric History | Safety Set |
| Listing 16.2.4.7 | Pregnancy Test Results | Safety Set |
| Listing 16.2.4.8 | Inclusion/Exclusion Criteria Failures | Safety Set |
| Listing I 6.2.4.9 | Eligibility Check | Safety Set |
| Listing 16.2.4.10 | Bag Search and Cigarette Collection | Safety Set |




| Listing 16.2.5.1 | Plasma Cytisine Concentration Data | Safety Set |
|---|---|---|
| Listing 16.2.5.2 | Urine Cytisine Concentration Data | Safety Set |
| Listing 16.2.5.3 | Individual Derived Plasma and Urine Cytisine Pharmacokinetic Parameters | Safety Set |
| Figure 16.2.5.1 | Individual Plasma Cytisine Concentration-Time Curves on a Linear Scale | Safety Set |
| Figure 16.2.5.2 | Individual Plasma Cytisine Concentration-Time Curves on a Semi-Logarithmic Scale | Safety Set |

## 16.2.6 Efficacy

Not applicable.

## 16.2.7 Adverse Events

| Listing 16.2.7.1 Adverse Events Safety Set |
|--------------------------------------------|
|--------------------------------------------|

## 16.2.8 Individual Laboratory Safety Measurements

| Listing 16.2.8.1 | Biochemistry Data | Safety Set |
|------------------|-----------------------|------------|
| Listing 16.2.8.2 | Haematology Data | Safety Set |
| Listing 16.2.8.3 | Urinalysis Data | Safety Set |
| Listing 16.2.8.4 | Microscopy Data | Safety Set |
| Listing 16.2.8.5 | Other Laboratory Data | Safety Set |

## 16.2.9 Vital Signs

| 11.11.12.00.1 | V/: 1 C: D : | |
|------------------|------------------|------------|
| Listing 16.2.9.1 | Vital Signs Data | Safety Set |
| LISCHIE 10.2.7.1 | Vical Oigns Data | Salety Set |
| _ | • | · |

# 16.2.10 Physical Examination

| Listing 16.2.10.1 Physical Examination Data | Safety Set |
|---------------------------------------------|------------|
|---------------------------------------------|------------|

#### 16.2.11 ECG

| Listing 16.2.11.1 | 12-Lead ECG Data | Safety Set |
|-------------------|------------------|------------|






## 16.2.12 Prior and Concomitant Medication

Listing 16.2.12.1 Prior and Concomitant Medication Use Safety Set

## 16.2.13 Pharmacodynamics

Not applicable.






# 15 SHELLS FOR TABLES, FIGURES AND LISTINGS




Achieve Life Sciences, Inc.: ACH-CYT-07 Statistical Analysis Plan










Achieve Life Sciences, Inc.: ACH-CYT-07 Statistical Analysis Plan


Achieve Life Sciences, Inc.: ACH-CYT-07 Statistical Analysis Plan




Achieve Life Sciences, Inc.: ACH-CYT-07 Statistical Analysis Plan ACH-CYT-07
























































































































































## **16 APPENDICES**

## 16.1 NORMAL RANGES

## Vital Signs Normal Ranges:

| Parameter | Normal Range | Units |
|--------------------------|--------------|------------------------|
| Pulse Rate | 40-100 | Beats per minute (bpm) |
| Systolic Blood Pressure | 90-140 | mmHg |
| Diastolic Blood Pressure | 50-90 | mmHg |
| Respiratory Rate | 12-18 | Breaths per minute |
| Oral Temperature | 35.0-37.5 | Degrees Celsius (°C) |
| Pulse Oximetry | 94-100 | % |

## 12-Lead ECG Normal Ranges:

| Parameter | Normal Range | Units |
|-------------------------------------|--------------|------------------------|
| Heart Rate | 40-100 | Beats per minute (bpm) |
| PR Interval | 120-220 | mSec |
| QRS Width | 70-120 | mSec |
| QT Interval | N/a | N/a |
| QTc Interval (=QTcF) (Fridericia's) | 350-450 | mSec |
